CLINICAL TRIAL: NCT05927727
Title: Benign-Malign Differentiation Of Axillary Lymph Nodes: The Role Of Superb Microvascular Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Oguzhan Tokur, Principal Investigator, Ankara Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Oguzhan Tokur
Record Dates: First submitted 2022-11-28; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Diagnosis; Axilla; Breast
Keywords: Axilla; Lymph node; Ultrasound; Doppler; Malignancy; SMI; PDUS
MeSH Terms: conditions — Disease; Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Malign Group (Active Comparator): The group includes patients who have malignant axillary lymph nodes which are proven by biopsy
  Interventions: Diagnostic Test: Ultrasound and biyopsy
- Benign Group (Active Comparator): The group includes patients who have benign axillary lymph nodes which are proven either by biopsy or follow-up
  Interventions: Diagnostic Test: Ultrasound and biyopsy

INTERVENTIONS:
Diagnostic Test: Ultrasound and biyopsy — Each participant has undergone to ultrasound and biopsy procedure if they have suspicious lymph node in axillar region

SUMMARY:
102 patients who have suspicious ALNs were included in our prospective study, which was approved by a tertiary health care facility ethics committee. Each suspicious lymph nodes (LNs) were examined with PDUS and SMI in terms of distribution, appearance and number of vascular structures and the still images were stored. Subsequently, imaging findings were re-evaluated after histopathological or follow-up results and were compared between benign and malign groups. In addition, we revealed the diagnostic perfomance of using the each possible combination of these features in PDUS and SMI. Finally, two radiologists with 22 years and 4 years of experience analyzed the images and interobserver agreement was assessed

DETAILED DESCRIPTION:
MATERIAL AND METHOD Patient The hospital's ethics committee approved this single-center prospective study (E-93471371-514.10). 139 female patients, ages 18 to 74, who had suspicious lymph nodes in the axilla during a breast ultrasound examination at our clinic between April 2021 and April 2022 were included in the study. 20 patients did not come back for follow-ups, 4 patients' ultrasonographic images were not sufficient diagnostic quality, and 13 patients were excluded from the study because the biopsy result was not diagnostic and the patient did not undergo re-biopsy. As a result, 108 lymph nodes from 102 patients were included in the study, and 37 patients were excluded.

Patients who were male, under the age of 18, underwent axillary lymph node dissection, had active infection in the axillary region, were diagnosed with histopathologically confirmed axillary lymph node metastasis, had received known chemotherapy or radiotherapy to the axillary region, or did not sign the informed consent form were excluded from the study. Patients who had their pathology results unavailable or who later decided not to participate in the study were also excluded.

Ultrasonographic Evaluation Suspicious axillary lymph nodes in the patients included in the study were evaluated with Toshiba Aplio a (Toshiba Medical Systems Corporation, Tokyo, Japan) ultrasound (US) device and 14-18 MHz high frequency linear probe. Gray scale US, PDUS and SMI images of the lymph nodes were stored. PRF and gain settings were adjusted to prevent from artifacts and to obtain the highest amount of signal while images were taken. In both Doppler methods, these parameters remained unchanged. The routine examination time for each patient extended 1-2 minutes by the SMI evaluation. At the end of the evaluation, a histological assessment using a 21G fine needle aspiration (FNA) biopsy or core biopsy (16-18G) from the relevant lymph nodes, or follow-up with US was performed, depending on the clinical suspicion. Any lymph nodes that regressed or disappeared throughout the US follow-up period of 1-3 months were considered benign. The lymph nodes that remained stable or progressed were evaluated through histopathological sampling. In case of non-diagnostic biopsy, patients were recalled and FNA/core biopsy was repeated. Cytology and pathology specimens were evaluated by a pathologist with at least 10 years of experience. Before the histopathological diagnosis, all patients were prospectively evaluated with ultrasonography by a radiologist blinded to the patient's clinic and history, and images were taken. After the pathology results, PDUS and SMI images were re-evaluated and the findings were compared with each other and pathology results. Finally, two radiologists with 22 years and 4 years of experience evaluated the images in terms of separately determined features without knowing the patient's clinical information and pathology result. The results were compared with each other in order to assess interobserver agreement.

Both PDUS and SMI assessed vascular patterns based on the number of internal vessels, the distribution (avascular/central/peripheral/mixed) and appearance (normal, dysplasic, avascular) of internal vessels. On SMI, both monochrome (mSMI) and color (cSMI) images were assessed. If there was diffuse cortical thickening of the lymph node, the entire cortex was included the images. Likewise if there was an asymmetric cortical thickening, images focused on that part.

Cortical flow signals were taken into account while internal vascularity was quantified. The lymph nodes with no vascular signals in the cortex were classified as avascular, the nodes with peripheral vascular signals as peripheral, the nodes with vascular signals extending from the hilus to the cortex as central, and the nodes with vascular signals in both the periphery and the central as mixed. To evaluate the morphology of the vessels, the signals with smooth, symmetrical hilar extension were considered as normal, the eccentric signals were identified as diplasic, and the lymph nodes without a signal were regarded as avascular.

Statistical Analysis In the study, mean and standard deviation were used for continuous variables, while frequency and percentage values were used when specifying categorical variables. The Kolmogorov-Smirnov and Shapiro Wilk test was used to evaluate the homogeneity of the patient distribution. Student t-test and Mann Whitney U test were used for continuous variables. Chi-square test or Fisher's exact chi-square test was used to evaluate categorical features In order to evaluate the diagnostic performance of each investigated feature of Doppler methods in the differentiation of benign and malignant lymph nodes, the area under the curve (AUC) was calculated separately by receiver operating characteristic (ROC) analysis, depending on whether they were used individually or together. Logistic regression analysis was used to determine the significance value when the features were used together. In addition, sensitivity, specificity, positive predictive value(PPV), negative predictive value (NPV) and accuracy of each method were evaluated.

The Kohen Kappa test was used for categorical features in both SMI and PDUS to assess interobserver agreement. Intragroup correlation coefficient test was used to compare vascular numbers. Chi-square test or Fisher's exact chi-square test was used to evaluate vascular properties between benign and malignant categories after consensus.

All statistical analyses was performed with SPSS version 25.0 (IBM Corp. Armonk, NY: USA. Released 2017). P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Female gender,
* Sign the informed consent form,
* No history of axillary lymph node metastasis histopathologically,
* No history of received chemotherapy or radiotherapy to the axillary region before,
* No history of axillary lymph node dissection
* No active infection in the axillary region.

Exclusion Criteria:

* Male patients,
* Under the age of 18,
* No history of histopathologically confirmed axillary lymph node metastasis,
* No history of chemotherapy or radiotherapy to the axillary region,
* Refuse to sign informed consent form
* Unavailable pathological result

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 102 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
The number of vascularity in both benign and malignant axillary lymph nodes | Up to three months
  The number of vascularity in axillary lymph nodes are assessed via inspection of the images of Superb Microvascular Imaging and Power Doppler Ultrasound by observers. Countable vascular signals are noted for each lymph nodes
The distribution of vessels in both benign and malignant axillary lymph nodes | Up to three months
  Vascular distributions in axillary lymph nodes are assessed via inspection of the images of Superb Microvascular Imaging and Power Doppler Ultrasound by observers and are categorized as avascular, central, peripheral and mix.
The appearance of vessels in both benign and malignant axillary lymph nodes | Up to three months
  Vascular appearance in axillary lymph nodes are assessed via inspection of the images of Superb Microvascular Imaging and Power Doppler Ultrasound by observers and are categorized as normal/central,eccentric, avascular.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Seher Oztekin, Assoc. Prof., Study Director — Ankara Education and Research Hospital
Locations (1):
- Ankara Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurt SA, Eryurekli AE, Kayadibi Y, Samanci C, Velidedeoglu M, Onur I, Arslan S, Taskin F. Diagnostic Performance of Superb Microvascular Imaging in Differentiating Benign and Malignant Axillary Lymph Nodes. Ultrasound Q. 2023 Jun 1;39(2):74-80. doi: 10.1097/RUQ.0000000000000617. PMID 35943392
- [Background] Uslu H, Tosun M. The benefit of superb microvascular imaging and shear wave elastography in differentiating metastatic axillary lymphadenopathy from lymphadenitis. Clin Breast Cancer. 2022 Aug;22(6):515-520. doi: 10.1016/j.clbc.2022.03.008. Epub 2022 May 6. PMID 35644841
- [Background] Zhu AQ, Li XL, An LW, Guo LH, Fu HJ, Sun LP, Xu HX. Predicting Axillary Lymph Node Metastasis in Patients With Breast Invasive Ductal Carcinoma With Negative Axillary Ultrasound Results Using Conventional Ultrasound and Contrast-Enhanced Ultrasound. J Ultrasound Med. 2020 Oct;39(10):2059-2070. doi: 10.1002/jum.15314. Epub 2020 May 5. PMID 32367518
- [Background] Bian J, Zhang J, Hou X. Diagnostic accuracy of ultrasound shear wave elastography combined with superb microvascular imaging for breast tumors: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2021 Jun 25;100(25):e26262. doi: 10.1097/MD.0000000000026262. PMID 34160389
- [Background] Kijima Y, Yoshinaka H, Hirata M, Mizoguchi T, Ishigami S, Nakajo A, Arima H, Ueno S, Natsugoe S. Number of Axillary Lymph Node Metastases Determined by Preoperative Ultrasound is Related to Prognosis in Patients with Breast Cancer. Cancers (Basel). 2010 Feb 4;2(1):20-31. doi: 10.3390/cancers2010020. PMID 24281030
- [Background] Yang WT, Chang J, Metreweli C. Patients with breast cancer: differences in color Doppler flow and gray-scale US features of benign and malignant axillary lymph nodes. Radiology. 2000 May;215(2):568-73. doi: 10.1148/radiology.215.2.r00ap20568. PMID 10796941
- [Background] Fu Z, Zhang J, Lu Y, Wang S, Mo X, He Y, Wang C, Chen H. Clinical Applications of Superb Microvascular Imaging in the Superficial Tissues and Organs: A Systematic Review. Acad Radiol. 2021 May;28(5):694-703. doi: 10.1016/j.acra.2020.03.032. Epub 2020 May 5. PMID 32418782
- [Background] Ryoo I, Suh S, You SH, Seol HY. Usefulness of Microvascular Ultrasonography in Differentiating Metastatic Lymphadenopathy from Tuberculous Lymphadenitis. Ultrasound Med Biol. 2016 Sep;42(9):2189-95. doi: 10.1016/j.ultrasmedbio.2016.05.012. Epub 2016 Jun 25. PMID 27353493
- [Background] Esen G, Gurses B, Yilmaz MH, Ilvan S, Ulus S, Celik V, Farahmand M, Calay OO. Gray scale and power Doppler US in the preoperative evaluation of axillary metastases in breast cancer patients with no palpable lymph nodes. Eur Radiol. 2005 Jun;15(6):1215-23. doi: 10.1007/s00330-004-2605-9. Epub 2005 Feb 3. PMID 15690206
- [Background] Ying M, Ahuja A, Brook F. Accuracy of sonographic vascular features in differentiating different causes of cervical lymphadenopathy. Ultrasound Med Biol. 2004 Apr;30(4):441-7. doi: 10.1016/j.ultrasmedbio.2003.12.009. PMID 15121245
- [Result] Sim JK, Lee JY, Hong HS. Differentiation Between Malignant and Benign Lymph Nodes: Role of Superb Microvascular Imaging in the Evaluation of Cervical Lymph Nodes. J Ultrasound Med. 2019 Nov;38(11):3025-3036. doi: 10.1002/jum.15010. Epub 2019 Apr 3. PMID 30945325